CLINICAL TRIAL: NCT02783235
Title: Cervical Cancer Screening: Video-based Tutorials for Skills Development of ANMs/ASHAs/PHWs
Brief Title: Cervical Cancer Screening : Video Based Tutorials for ANMs/ASHAs/PHWs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Gauravi Ashish Mishra, Associate Professor Dept of Preventive Oncology, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TMH1605 Video Based Tutorials
Record Dates: First submitted 2016-05-16; First posted 2016-05-26 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Cervical Cancer
Keywords: VIA; Cervical Cancer; Training
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cervical cancer (Other): cervical cancer screening and training for ANMs/ASHAs/PHWs To develop video-based tutorials to train ANMs/ASHAs/PHWs in conducting cervical cancer related health education, screening for cervical cancers using VIA, collection of PAP smears and HPV samples.
  Interventions: Other: cervical cancer screening

INTERVENTIONS:
Other: cervical cancer screening — for 50 ANMs/ASHAs/PHWs/ in conducting cervical cancer related health education , screening for cervical cancers using VIA, collection of PAP smears and HPV samples.

SUMMARY:
This study aims at creating video-based tutorials for developing skills in performing cervical cancer screening using VIA for the Auxillary Nurse Midwives (ANMs), Accredited Social Health Activists (ASHAs) and Primary Health Workers (PHWs). Cervical cancer screening is mainly done by the following three methods: Visual inspection with acetic acid (VIA), Cervical Smear Cytology (PAP) and HPV DNA test. VIA is a low cost, low resource cervical cancer screening method and especially useful for low middle income countries (LMICs) like India.

We propose to develop video-based tutorials, such that the ANMs/ASHAs/PHWs could be trained in performing and interpreting VIA with the use of this tutorial. The ANMs/ASHAs/PHWs have important roles in delivering health in rural/ semi urban areas and they will be trained using this tutorial.

The video-based tutorials will be made according to the 'Spoken Tutorials' methodology, developed at IIT Bombay. Video-based Tutorials has given skills based training to over 2 lakh students in the past four years on IT based topics. The tutorials are made available online free of cost. They are designed to be used without the need of an expert being physically present.

DETAILED DESCRIPTION:
Aim of the study:

1. To develop video-based tutorials to train ANMs/ASHAs/PHWs in conducting cervical cancer related health education, screening for cervical cancers using VIA, collection of PAP smears and HPV samples.
2. To reduce the training time required by an expert to train ANMs/ASHA/PHWs as compared to the traditional training methods.
3. To evaluate the efficacy of the training tool by conducting a pre-test and post-test and practical test for lesion identification.
4. To assess the satisfaction levels of ANMs/ASHAs/PHWs for learning through video-based tutorials.

Methodology:

A. Creating the Tutorials

1) The video-based tutorials will be created with the help of domain experts, Content generators and Animators.

B. Conducting the Training

1. TMH will recruit Medical Social Workers and Health Workers to provide training to 50 ANMs/ASHAs/PHWs at their own centres.
2. The training will be staggered into different modules, and will be completed for each trainee over a period of approximately 3 months.

The investigators will also obtain images after due permissions, of the clinic, preparations for examination like arrangements of trolleys, preparation of dilute acetic acid, etc. and the cervical pictures/ videos of the patients before and after VIA after obtaining due consents (there will be no revealing of identity) to aid the animation and the tutorials.

The effectiveness of the tutorials will be checked by a pre- and post- tutorial assessment quiz.

Sample Size and power estimates:

For this study, sampling method is a convenience sample of 50 ANMs/ASHAs/PHWs attached to the TMC, District, Municipal Hospitals and PHCs who have not learned VIA based cervical cancer screening before.

Three MSWs will be appointed to co-ordinate with the respective officials of BMC, State Government, District hospitals etc. and explain the importance of the project.

The Social Workers will approach different BMC hospitals in Mumbai and PHCs and district hospitals around Mumbai to relieve their ANMs/ASHAs/PHWs to participate in this training. Newly recruited PHWs in the Preventive Oncology projects will also be enrolled for this training.

1. Pre training knowledge about various aspects of cervical cancer viz., causes, various cervical cancer screening techniques, steps required to perform VIA etc.
2. The satisfaction level and feed back of the trainees with the course provided.
3. Improvement in the Post training knowledge about various aspects of cervical cancer viz., causes, various cervical cancer screening techniques, steps required to perform VIA etc.

   These will be measured with the help of test scores. Each question in the test will have marks assigned to it based on difficulty level. (Easy 1 mark, Intermediate 2 marks, Hard 3 marks, Very hard 4 marks). The ANMs will be assigned marks depending on the number of correct responses.

   The ANMs will have to take the tests before the training, immediately after the training, and three months after the training is complete.

   The satisfaction level with the mode of teaching will be done on a survey based on a likert scale.
4. Ability to correctly identify a VIA positive lesion.

This will be measured based on marks they score during the tests and assignments, where they will do an image based diagnosis of 15 VIA cases. This will also be scored based on observation sessions they will have with a doctor who performs VIA on 10 patients. They will be assessed based on the number of correct identifications of VIA lesions.

Data entry and analysis:

Data entry will be done in IIT Bombay and in the Department of Preventive Oncology, Tata Memorial Hospital, using SPSS version 18. Checks for consistency, data safety and analysis will be carried out at regular intervals. Both descriptive and inferential statistics will be generated for describing variables under the study objectives.

Agreement of test scores, pre-training and post-training will be estimated using kappa statistics.

ELIGIBILITY:
Inclusion Criteria: ANMs /ASHAs/PHWs attached to the TMC, District Hospitals and PHCs who have not learned VIA based cervical cancer screening before.

Exclusion Criteria: ANMs /ASHAs/PHWs attached to the TMC, District Hospitals and PHCs who have learnt VIA based cervical cancer screening before.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in the Post training knowledge about cancer | 1 year
  Questionnaire: that will compare pre-training knowledge with post training and assess the improvement in the Post training knowledge about various aspects of cervical cancer viz., causes, various cervical cancer screening techniques, steps required to perform VIA etc.
  These will be measured with the help of test scores. Each question in the test will have marks assigned to it based on difficulty level. (Easy 1 mark, Intermediate 2 marks, Hard 3 marks, Very hard 4 marks). The ANMs will be assigned marks depending on the number of correct responses.
  The ANMs will have to take the tests before the training, immediately after the training, and three months after the training is complete.

SECONDARY OUTCOMES:
Satisfaction to the video based tutorials | 1 year
  Questionnaire: that will assess the satisfaction level and feed back of the trainees with the course provided.
  The satisfaction level with the mode of teaching will be done on a survey based on a likert scale.

OTHER OUTCOMES:
Clinical skills development | 1 year
  Scores will be assigned and the ability to correctly identify a VIA positive lesion will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Gauravi A Mishra, MD, Principal Investigator — Tata Memorial Hospital, Mumbai.; Gauravi A Mishra, MD, Principal Investigator — ata Memorial Hospital, Mumbai.
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
Data entry will be done in IIT Bombay and in the Department of Preventive Oncology, Tata Memorial Hospital, using SPSS version 18.

REFERENCES:
- See also: Tata Memorial Centre, Mumbai Official website — http://tmc.gov.in